CLINICAL TRIAL: NCT01680666
Title: A Prospective Randomized Trial of Ultrasound Versus Landmark Guided Central Venous Access in Children
Brief Title: A Prospective Trial of Ultrasound Versus Landmark Guided Central Venous Access in the Pediatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Matias Bruzoni, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-8943
Record Dates: First submitted 2012-08-28; First posted 2012-09-07 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Need for Central Venous Access
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- landmark guided (Active Comparator): central line placement
  Interventions: Procedure: central line placement
- ultrasound guided (Active Comparator): central line placement
  Interventions: Procedure: central line placement; Device: Ultrasound

INTERVENTIONS:
Procedure: central line placement — central line placement
Device: Ultrasound — Ultrasound guided central venous access
  Other Names: Sonosite, Bothel, WA; Aloka, Wallingford, CT
  Arms: ultrasound guided

SUMMARY:
The investigators hypothesized that, in children undergoing venous cannulation for central line placement by pediatric surgeons, ultrasound-guided cannulation leads to an increase in successful venous cannulation at first attempt compared to landmark guided cannulation.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 0 and 18 years undergoing tunneled central venous line placement under general anesthesia

Exclusion Criteria:

* Preoperative proof of non-patency of central veins
* coagulopathy
* access site surgeon

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - Children's Mercy Hospital, Kansas City, Missouri

REFERENCES:
- [Result] Bruzoni M, Slater BJ, Wall J, St Peter SD, Dutta S. A prospective randomized trial of ultrasound- vs landmark-guided central venous access in the pediatric population. J Am Coll Surg. 2013 May;216(5):939-43. doi: 10.1016/j.jamcollsurg.2013.01.054. Epub 2013 Mar 7. PMID 23478546

RESULTS

PARTICIPANT FLOW:
Groups:
- Landmark Guided: In the landmark technique, the subclavian vein or the internal jugular vein on either side was chosen for access depending on surgeon's preference. An infraclavicular approach was used for the subclavian vein, and an anterior approach was used for the internal jugular vein. If venous flash could not be achieved after three attempts on the initial chosen site using the landmark technique, the study was terminated and the surgeon was free to use either ultrasound or landmark at any other site. A single pass of the needle was defined as a single episode of needle advancement and withdrawal. A second pass occurred if the needle was re-advanced or removed and reinserted. A failed attempt was recorded if aspiration resulted in no venous flash, arterial puncture (bright red blood, pulsatile flow), or air.
- Ultrasound Guided: In the ultrasound-guided group, the internal jugular vein on either side was accessed depending on surgeon's preference. An ultrasound console with a linear 11 Hz probe was used. The patient was then put into Trendelenburg position. The head was positioned away from the insertion side. The ultrasound probe was placed at the apex of the triangle formed between the two heads of the sternocleidomastoid muscle and the clavicle. The internal jugular vein and common carotid artery were visualized, with the vein identified by its larger size, relative anatomic position, and compressibility. After a flashback of dark venous blood was noted in the syringe, the standard Seldinger technique was followed for the catheter insertion. After 3 failed attempts using the ultrasound at the specified site, the surgeon was free to further attempts using landmark or ultrasound approaches at any other site.
Period: Overall Study
Arm/Group | Landmark Guided | Ultrasound Guided
Started | 84 | 66
Completed | 84 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Landmark Guided | Ultrasound Guided | Total
Number analyzed (Participants) | 84 | 66 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 84 | 66 | 150
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 8 [0 to 18] | 5 [0 to 18] | 7 [0 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 23 | 54
  Male | 53 | 43 | 96
Region of Enrollment [Number; unit: participants]
  United States | 84 | 66 | 150

OUTCOME MEASURES:

1. Primary Outcome: Success of Central Venous Cannulation at First Attempt
Description: The count (%) of patients with successful central venous cannulation at first attempt is reported.
Time Frame: Up to 410 seconds
Measure: Count of Participants; unit: Participants
Groups:
- Landmark Technique: In the landmark technique, the subclavian vein or the internal jugular vein on either side was chosen for access depending on surgeon's preference. An infraclavicular approach was used for the subclavian vein, and an anterior approach was used for the internal jugular vein. If venous flash could not be achieved after three attempts on the initial chosen site using the landmark technique, the study was terminated and the surgeon was free to use either ultrasound or landmark at any other site. A single pass of the needle was defined as a single episode of needle advancement and withdrawal. A second pass occurred if the needle was re-advanced or removed and reinserted. A failed attempt was recorded if aspiration resulted in no venous flash, arterial puncture (bright red blood, pulsatile flow), or air.
Arm/Group | Landmark Technique | Ultrasound Guided
Number analyzed (Participants) | 84 | 66
Participants | 38 | 43

2. Secondary Outcome: Success of Central Venous Cannulation Within First Three Attempts
Description: The count (%) of patients with successful central venous cannulation within the first three attempts is reported.
Time Frame: Up to 410 seconds
Measure: Count of Participants; unit: Participants
Arm/Group | Landmark Guided | Ultrasound Guided
Number analyzed (Participants) | 84 | 66
Participants | 62 | 63

3. Secondary Outcome: Patients With Arterial Punctures
Description: The count (%) of patients with arterial punctures is presented.
Time Frame: Up to 410 seconds
Measure: Count of Participants; unit: Participants
Arm/Group | Landmark Guided | Ultrasound Guided
Number analyzed (Participants) | 84 | 66
Participants | 7 | 3

4. Secondary Outcome: Patients With Complications
Description: The count (%) of patients with complications (including hemothorax, hematoma, pneumothorax, or catheter malposition) is presented.
Time Frame: Up to 410 seconds
Measure: Count of Participants; unit: Participants
Arm/Group | Landmark Guided | Ultrasound Guided
Number analyzed (Participants) | 84 | 66
Participants | 4 | 3

5. Secondary Outcome: Time to Successful Cannulation
Time Frame: Up to 410 seconds
Measure: Mean (Full Range); unit: seconds
Arm/Group | Landmark Guided | Ultrasound Guided
Number analyzed (Participants) | 84 | 66
seconds | 42 [4 to 410] | 33 [2 to 220]

ADVERSE EVENTS:
Time Frame: Up to 410 seconds
Description: Per protocol, procedure-related complications were reported as adverse events
Arm/Group | Landmark Guided | Ultrasound Guided
Serious Adverse Events (participants affected / at risk) | 11/84 | 6/66
Other Adverse Events (participants affected / at risk) | 0/84 | 0/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Landmark Guided (N=84) | Ultrasound Guided (N=66)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hematoma (nonexpanding) (Vascular disorders) | 2 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Arterial puncture (Vascular disorders) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No